CLINICAL TRIAL: NCT05806710
Title: Safety and Acceptance of GourMed© Prepackaged Nutritional Products in the Elderly Dysphagic Patient: MODiet Project
Acronym: MODiet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: INRCA_002_2023
Record Dates: First submitted 2023-03-27; First posted 2023-04-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-03

CONDITIONS: Dysphagia
Keywords: dysphagia; diet; elderly subjects
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dysphagic subjects (Experimental): elderly patients with dysphagia
  Interventions: Dietary Supplement: GourMed© meal

INTERVENTIONS:
Dietary Supplement: GourMed© meal — patients receive GourMed© meal as lunch for 7 consecutive days

SUMMARY:
The aim of the MoDiet study is to evaluate the usefulness of the GourMed© prepackaged diet in guaranteeing a safe, compliant and effective diet satisfying the nutritional needs of the elderly dysphagic patient.

DETAILED DESCRIPTION:
The objective of the MoDiet study is to evaluate the usefulness of the GourMed© (MedicAir Food srl, Milano, Italy) prepackaged diet in guaranteeing a safe, compliant and effective diet satisfying the nutritional needs of the elderly dysphagic patient.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years and over
* Gugging Swallowing Screen ranging 10-20;

Exclusion Criteria:

* known or suspected intolerance to any ingredient
* taking other prepackaged products for dysphagia
* creatinine ≥1,5 mg/dl

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-03-11 (Estimated); Study Completion 2024-03-11 (Estimated)

PRIMARY OUTCOMES:
safety of GourMed© meal | during each GourMed© meal (up to day 7)
  The safety of GourMed© meal is monitoring by the registration of the following events:
  * Appearance of coughing and/or changes in the tone of voice immediately after or within 1-2 minutes of swallowing a bite;
  * Spill of food from the nose;
  * Prolonged management of the bolus in the oral cavity
  * Appearance of red or cyanotic color on the face
  * Occurrence of allergic skin reactions
  * Appearance of breathing difficulties
  * Onset of fever
  * Appearance of nausea, vomiting or diarrhea.

SECONDARY OUTCOMES:
evaluate the amount of GourMet© meal consumed | after each GourMed© meal (up to day 7)
  The amount of GourMet© meal is recorded to verify that the patient's nutritional needs are met

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS INRCA Hospital, Casatenovo, Lecco
  - Ospedale Mandic, Merate, Lecco
  - IRCCS INRCA Hospital, Ancona